CLINICAL TRIAL: NCT05186779
Title: Maternal and Newborn Safety Profile of Progestogens in EARLY Pregnancy
Acronym: PEARLY
Status: Terminated | Type: Observational
Why Stopped: Challenges in recruiting patients
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Abbott Products Operations AG (Unknown)
Responsible Party: Principal Investigator, Clare Barnett, MBBS (Hons) MPH, Dr. Clare Barnett, Center for Epidemiology and Health Research, Germany
Other Study IDs: DYDR5007
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Early Pregnancy Bleeding; Recurrent Pregnancy Loss
MeSH Terms: interventions — Progestins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Early Pregnancy Bleeding/Recurrent Pregnancy loss
  Interventions: Drug: Progestagen
- Cohort B: IVF/ART
  Interventions: Drug: Progestagen

INTERVENTIONS:
Drug: Progestagen — Subjects receiving treatment with any progestogen, including dydrogesterone, or other treatment in the first trimester of pregnancy following; (Cohort A) a diagnosis of early bleeding in pregnancy or recurrent pregnancy loss, or (Cohort B) following IVF/ART embryo transfer
  Other Names: Any other treatment for the indication as per cohort A or cohort B

SUMMARY:
This multinational, prospective, active surveillance, registry study following two cohorts will include study participants who are pregnant and seeking any type of medical treatment, including dydrogesterone and other progestogens, for either (A) recurrent pregnancy loss and/or bleeding in early pregnancy or (B) as In-Vitro Fertilization (IVF)/Assissted Reproductive Technology (ART) support. Pregnant women not taking progestogen and are advised an alternative non-medical treatment, in the context of bleeding in early pregnancy, recurrent pregnancy loss, or undergoing natural cycle frozen embryo transfer (NC-FET) can also be included in this study. Eligible study participants will be recruited via an international network of prescribing Health Care Practitioners (HCPs) in China, Turkey, and Russia with the aim to collect data related to maternal safety and newborn safety in women prescribed progestogens during early pregnancy. Study participants will be followed from early pregnancy until 6 - 12 weeks after giving birth. All malformations will be captured via direct contacts with the study participants. Study participants will be sent online questionnaires via the electronic Patient Reported Outcomes (ePRO) solution provided by MediData. Major malformations reported by the study participants will be validated by ZEG Berlin via relevant source documents and if necessary, via contacting the treating HCPs. The total study duration is planned for approximately 4 years including recruitment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who wish to sustain their pregnancy
* Women who have tested positive (blood or urine) for pregnancy in the first trimester
* treated with progestogens or any alternative treatment for early bleeding in pregnancy with evidence of an intrauterine pregnancy / unexplained recurrent OR pregnancy loss (with ≥ 2 previous pregnancy losses) with evidence of an intrauterine pregnancy OR having undergone IVF/ ART embryo transfer and taking progestogen for luteal phase support (LPS), with evidence of an intrauterine pregnancy
* Signed informed consent, allowing consent to contact all treating, or diagnosing HCP
* Able and willing to read and comprehend written instructions; comprehend and complete the questionnaires required by the protocol

Exclusion Criteria:

* Serious disease or disease requiring teratogenic treatment (e.g., Lupus Erythematosus, Multiple Sclerosis, cancer)
* Multifetal pregnancy
* More than four (4) previous IVF embryo transfers
* Previous exposure to dydrogesterone in index pregnancy
* Documented substance abuse
* Treatment with hormones which are known to cause malformations
* Participation in an observational study that might, in the recruiting HCP's opinion, influence the assessment for the current study
* Participation in a randomized clinical trial in the last 3 months
* Previous enrollment in the PEARLY study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects receiving treatment with any progestogen, including dydrogesterone, or other treatment in the first trimester of pregnancy following; (A) a diagnosis of early bleeding in pregnancy or recurrent pregnancy loss,or (B) following IVF/ART embryo transfer will be eligible to be enrolled. Subjects can be screened for the study only after an informed decision for dydrogesterone or alternative treatment has been made by the subject and the recruiting HCP. Indication and contraindications according to the local market authorization/ summary of product characteristics (SmPC) should be carefully considered by the HCP.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
the rate of major malformations in fetus by indication and by exposure to progestogens during the first trimester of pregnancy, with an emphasis on dydrogesterone versus non-dydrogesterone treatments. | at approximately 24 weeks of pregnancy
the rate of major malformations in newborns by indication and by exposure to progestogens during the first trimester of pregnancy, with an emphasis on dydrogesterone versus non-dydrogesterone treatments. | at 6-12 weeks after the initial estimated date of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Clare Barnet, Principal Investigator — ZEG
Locations (1):
- Center for Epidemiology and Health Research Berlin, Berlin, Germany